CLINICAL TRIAL: NCT02516384
Title: Fecal Microbiota Transplantation (FMT) in the Management of Ulcerative Colitis (UC)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1404014982
Record Dates: First submitted 2015-07-29; First posted 2015-08-05 (Estimated); Last update posted 2018-02-22 (Actual); Status verified 2018-02

CONDITIONS: Ulcerative Colitis
Keywords: Fecal Microbiota Transplantation; Ulcerative Colitis
MeSH Terms: conditions — Colitis, Ulcerative | interventions — Fecal Microbiota Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Fecal Microbiota Transplantation (Experimental): Individuals with Ulcerative Colitis will undergo a fecal microbiota transplantation.
  Interventions: Biological: Fecal Microbiota Transplantation

INTERVENTIONS:
Biological: Fecal Microbiota Transplantation — We will use fecal microbiota transplantation (FMT), with fecal material obtained from OpenBiome or donor directed, to assess safety (as primary outcome) and efficacy (as secondary outcome) in adult (>18 year old) patients with active ulcerative colitis (UC).

SUMMARY:
Inflammatory bowel disease is a condition caused by gastrointestinal immune system dysregulation and affected by both genetic and environmental factors. Differences in intestinal bacteria exist between IBD patients and healthy controls, but the role of intestinal bacteria in the development and treatment of IBD remains largely unknown. Fecal microbiota transplantation (FMT) is the transfer of gastrointestinal bacteria from a healthy donor to a patient with altered microbial diversity with the intent of restoring a normal bacterial balance. Most studies focus on its use in treating Clostridium difficile (CDI), an infection characterized by dysbiosis. Given the role of dysbiosis in IBD, the investigators hypothesize that FMT may be beneficial in IBD. The purpose of this study is to prospectively examine the safety of FMT in the management of ulcerative colitis (UC).

DETAILED DESCRIPTION:
Ulcerative colitis (UC) is a chronic inflammatory bowel disease (IBD) with significant morbidity and mortality. Current therapies remain limited by side effects and loss of response over time, and there is an ongoing need for new therapies. Fecal microbiota transplantation (FMT), which has proven to be safe and effective in the management of Clostridium difficile infection (CDI) has been proposed as a therapy for UC. There have been studies examining the role of FMT in UC, but they have shown mixed results, and have not examined the underlying immunologic and microbial changes to explain how and why FMT works from specific donors and in certain recipients. Furthermore, no studies have examined the long-term safety of FMT in patients with UC. This proposal aims to examine: (a) the short- and long-term safety of FMT in patients with UC, (b) the efficacy of FMT as a therapy for mild-moderate UC, and (c) the microbial and immunologic changes that occur after FMT, to help understand how and why it works in this group of patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients with biopsy proven ulcerative colitis (UC), including those with inadequately controlled UC (flare) as defined by failure of standard medical therapy, steroid-dependence, and/or need for escalation of medical care as determined by severity index (Mayo Score), endoscopic or histologic study, and/or medical provider
* Have active disease, defined with a Mayo Score > 3 and Mayo endoscopic subscore >1
* Subjects whom the investigator believes can and will comply with the requirements of the protocol
* Able to provide informed written consent.

Exclusion Criteria:

* Biopsy-proven Crohn's disease or indeterminate colitis
* Acute abdomen or other clinical emergencies requiring emergent management (for example: stricture, bowel obstruction, perforation and/or abscess)
* Primary sclerosing cholangitis (PSC)
* Pregnancy
* Concurrent Clostridium difficile infection or other known infection
* Prior history of fecal microbiota transplantation
* Other causes of diarrhea, including but not limited to tube feeds and medications (for example, kayaxelate, metformin, lactulose, laxatives, magnesium)
* Major congenital defects
* Subjects with recent malignancy in the last 5 years, excluding non-melanoma skin malignancies
* Anaphylactic reactions to any foods
* Any antibiotic use within the last 3 months
* Subject having any other condition that, in the opinion of the investigator, would jeopardize the safety or rights of the participant participating in the study, would make it unlikely for the participant to complete the study, or would confound the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2016-10-01 (Actual); Primary Completion 2016-12-31 (Actual); Study Completion 2017-01-31 (Actual)

PRIMARY OUTCOMES:
Safety post-FMT as determined by interview for adverse events | 36 months post-FMT
  Patient information regarding adverse events and safety of FMT for UC will be collected throughout the study period, including day 0, weeks 1, 2, 4, 6, 12 24, and then every 6 months until 36 months post-FMT. Throughout the study period, patients will be assessed for safety with questions regarding general well-being (such as "how have you been feeling?"), as well as specific questions to evaluate for occurrence of adverse events. Patients will also be questioned regarding stool form and frequency, presence of abdominal pain, fevers and subjective well-being.

SECONDARY OUTCOMES:
Clinical remission | 2, 4 and 12 weeks post fecal microbiota transplantation
  Defined by Mayo score ≤ 2 without any subscore >1, and Mayo endoscopic subscore 0-1
Clinical Response | 2, 4 and 12 weeks post fecal microbiota transplantation
  Defined by decrease in Mayo score by 3 points, decrease in bleeding subscore by 1, or absolute subscore of 0-1
Progression of disease defined by initiation of anti-TNF agents | 2, 4 and 12 weeks post fecal microbiota transplantation
  Initiation of anti-TNF agents (such as infliximab, adalimumab, certolizumab), vedolizumab, steroids. Includes time gap until additional agents are started
Progression of disease defined by increase in dosages of current UC medications | 2, 4 and 12 weeks post fecal microbiota transplantation
  Increase in dosages of current ulcerative colitis specific medications
Progression of disease defined by time to colectomy | up to three year follow-up period post fecal microbiota transplantation
  Time to colectomy rates and increase in time to colectomy
Death secondary to UC | Anytime during the three year follow-up period post fecal microbiota transplantation
  Time to death secondary to ulcerative colitis
Progression of disease defined by clinical flare | 2, 4 and 12 weeks post fecal microbiota transplantation
  Time to next flare
Microbial changes | 0, 2 and 4 weeks post fecal microbiota transplantation
  - Alterations in microbial profiles as defined by sequence of genetic material from fecal material.
Immunological changes | 0, 2 and 4 weeks post fecal microbiota transplantation
  - Alterations in immune cell function as defined by RNA sequencing and flow cytometry

CONTACTS AND LOCATIONS:
Overall Officials: Carl V Crawford, MD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Cornell Medical College, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Damman CJ, Miller SI, Surawicz CM, Zisman TL. The microbiome and inflammatory bowel disease: is there a therapeutic role for fecal microbiota transplantation? Am J Gastroenterol. 2012 Oct;107(10):1452-9. doi: 10.1038/ajg.2012.93. PMID 23034604
- [Background] Hanauer SB. Inflammatory bowel disease: epidemiology, pathogenesis, and therapeutic opportunities. Inflamm Bowel Dis. 2006 Jan;12 Suppl 1:S3-9. doi: 10.1097/01.mib.0000195385.19268.68. PMID 16378007
- [Background] Sartor RB, Muehlbauer M. Microbial host interactions in IBD: implications for pathogenesis and therapy. Curr Gastroenterol Rep. 2007 Dec;9(6):497-507. doi: 10.1007/s11894-007-0066-4. PMID 18377803
- [Background] Loftus EV Jr. Clinical epidemiology of inflammatory bowel disease: Incidence, prevalence, and environmental influences. Gastroenterology. 2004 May;126(6):1504-17. doi: 10.1053/j.gastro.2004.01.063. PMID 15168363
- [Background] Kunde S, Pham A, Bonczyk S, Crumb T, Duba M, Conrad H Jr, Cloney D, Kugathasan S. Safety, tolerability, and clinical response after fecal transplantation in children and young adults with ulcerative colitis. J Pediatr Gastroenterol Nutr. 2013 Jun;56(6):597-601. doi: 10.1097/MPG.0b013e318292fa0d. PMID 23542823
- [Background] Bennet JD, Brinkman M. Treatment of ulcerative colitis by implantation of normal colonic flora. Lancet. 1989 Jan 21;1(8630):164. doi: 10.1016/s0140-6736(89)91183-5. No abstract available. PMID 2563083
- [Background] van Nood E, Vrieze A, Nieuwdorp M, Fuentes S, Zoetendal EG, de Vos WM, Visser CE, Kuijper EJ, Bartelsman JF, Tijssen JG, Speelman P, Dijkgraaf MG, Keller JJ. Duodenal infusion of donor feces for recurrent Clostridium difficile. N Engl J Med. 2013 Jan 31;368(5):407-15. doi: 10.1056/NEJMoa1205037. Epub 2013 Jan 16. PMID 23323867
- [Background] Borody TJ, Campbell J. Fecal microbiota transplantation: techniques, applications, and issues. Gastroenterol Clin North Am. 2012 Dec;41(4):781-803. doi: 10.1016/j.gtc.2012.08.008. PMID 23101687
- [Background] Nagalingam NA, Lynch SV. Role of the microbiota in inflammatory bowel diseases. Inflamm Bowel Dis. 2012 May;18(5):968-84. doi: 10.1002/ibd.21866. Epub 2011 Sep 20. PMID 21936031
- [Background] Vermeire S JM, Verbeke K, al e. Pilot study on the safety and efficacy of faecal microbiota transplantation in refractory crohn's disease. Gastroenterology 2012, 142:S360.
- [Background] Angelberger S LC, Gratzer C, al. e. Fecal transplantation in patients with moderately to severely chronic active ulcerative colitis (UC). ECCO Conference Abstracts 2012:P374
- [Background] Kump PK, Grochenig HP, Lackner S, Trajanoski S, Reicht G, Hoffmann KM, Deutschmann A, Wenzl HH, Petritsch W, Krejs GJ, Gorkiewicz G, Hogenauer C. Alteration of intestinal dysbiosis by fecal microbiota transplantation does not induce remission in patients with chronic active ulcerative colitis. Inflamm Bowel Dis. 2013 Sep;19(10):2155-65. doi: 10.1097/MIB.0b013e31829ea325. PMID 23899544
- [Background] Greenberg A AO, Shelton C, Brandt L. Long-term Follow-up Study of Fecal Microbiota Transplantation (FMT) for Inflammatory Bowel Disease (IBD). Am J Gastroenterol 2013, 108:S540.
- [Background] Brandt L AO, Greenberg A, et al. Safety of Fecal Microbiota Transplantation (FMT) in Immunocompromised (Ic) Patients with Inflammatory Bowel Disease (IBD). Am J Gastroenterol 2013, 108:S556.
- [Derived] Lima SF, Gogokhia L, Viladomiu M, Chou L, Putzel G, Jin WB, Pires S, Guo CJ, Gerardin Y, Crawford CV, Jacob V, Scherl E, Brown SE, Hambor J, Longman RS. Transferable Immunoglobulin A-Coated Odoribacter splanchnicus in Responders to Fecal Microbiota Transplantation for Ulcerative Colitis Limits Colonic Inflammation. Gastroenterology. 2022 Jan;162(1):166-178. doi: 10.1053/j.gastro.2021.09.061. Epub 2021 Oct 2. PMID 34606847